CLINICAL TRIAL: NCT06515821
Title: Multicentre Observational Study for the Data Collection, Development and Evaluation of the Performance of Novel CRC Screening and Diagnostic Methods ONCOSCREEN-CS
Brief Title: Multicentre Study for Data Collection, Development, and Evaluation of Novel CRC Screening and Diagnostic Methods
Status: Recruiting | Type: Observational
Sponsor: Firalis SA (Industry)
Collaborators: University Medical Center Mainz (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A01793-42
Record Dates: First submitted 2024-06-28; First posted 2024-07-23 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer
Keywords: early CRC detection; biomarkers; diagnostic tool; high risk subject; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Breath, Faeces, Buccal swab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- CRC Group: Subject has positive CRC diagnosis according to colonoscopy result
  Interventions: Diagnostic Test: ONCOSCREEN
- Control Group with risks and presence of polyps: Healthy individuals with recognized risk factors for CRC development defined by either heredity and/or obesity and/or smoking and/or excess alcohol consumption and/or hyperlipidaemia.
  Interventions: Diagnostic Test: ONCOSCREEN
- Control Group with risks and absence of polyps: Healthy individuals with recognized risk factors for CRC development defined by either heredity and/or obesity and/or smoking and/or excess alcohol consumption and/or hyperlipidaemia.
  Interventions: Diagnostic Test: ONCOSCREEN
- Control Group with no risks: Healthy individuals without any recognized risk factors for CRC development defined by either heredity and/or obesity and/or smoking and/or excess alcohol consumption and/or hyperlipidemia.
  Interventions: Diagnostic Test: ONCOSCREEN

INTERVENTIONS:
Diagnostic Test: ONCOSCREEN — Subjects samples will be tested with diagnostic tests.

SUMMARY:
The primary goal is to develop easy accessible diagnostic tools for high risk subjects for colon cancer in different European populations to improve early CRC detection. These CRC screening technologies would be low cost, breakthrough and of high sensitivity and specificity.

DETAILED DESCRIPTION:
Colorectal Cancer (CRC) is the third most commonly occurring cancer in men and the second most commonly occurring cancer in women. CRC can often be prevented through regular screening. Although colonoscopy-based screening programs result in a significant decrease in CRC incidence, the compliance rate for performing the required screening remains too low and not the desired one. Fecal Occult Blood Test (FOBT) is another widely used screening modality for CRC but have certain constraints, such as relatively low sensitivity and the need for multiple sampling (three) to reach full screening potential. The development of novel, more practical screening methods can effectively increase the screening rates for CRC through non-invasive, repeatable, cost-effective, easy-to-use, and patient-friendly procedures. This is of particular importance in different European societies and population subgroups, since an increase in the incidence of Early-Onset CRC is currently noticed, which is significantly associated with risk factors such as heredity, obesity, smoking, alcohol abuse, and hyperlipidemia.

Within this framework, ONCOSCREEN will develop a multi-tier diagnostic solution towards improved CRC screening. Furthermore, ONCOSCREEN will consider specific socio-economic determinants which increase the regional or national CRC risks, thus exploiting new solutions, particularly in younger high-risk individuals in European communities. For the validation of the developed solution, a clinical validation study (titled "ONCOSCREEN-CS") will be conducted to assess its effectiveness, sensitivity, and specificity in detecting CRC at an early stage. During the first phase of the study (ONCOSCREEN-CS-Phase A), the investigators will identify the different expression patterns of the four diagnostic solutions (ONCO-VOC, ONCO-CRISP, ONCO-NMR, ONCO-CTC) in CRC patients and healthy controls with high risk for CRC, and also initially estimate their sensitivity and specificity. During the second phase (ONCOSCREEN-CS-Phase B), the ONCOSCREEN solution will be clinically validated.

ELIGIBILITY:
Inclusion Criteria:

* CRC Group

  1. Signature of the informed consent indicating that the subject accepts to participate in the study and to comply with the requirements and restrictions inherent in this study.
  2. Subjects aged ≥18 years
  3. Subject is willing to undergo FOBT test, colonoscopy, and tissue biopsy
  4. Subject for whom the decision to perform a colonoscopy has been made by the treating physician
  5. Subject has positive CRC diagnosis according to colonoscopy result
  6. Covered by a Health Insurance System
  7. Subject is able to comply with all study procedures
* Control Group with risks and presence of polyps

  1. Signature of the informed consent indicating that the subject accepts to participate in the study and to comply with the requirements and restrictions inherent in this study.
  2. Subjects aged ≥18 years
  3. Otherwise healthy individuals with recognized risk factors for CRC development defined by either heredity and/or obesity and/or smoking and/or excess alcohol consumption and/or hyperlipidaemia.
  4. Subject be willing to undergo FOBT test, colonoscopy, and tissue biopsy
  5. Subject has negative CRC diagnosis according to colonoscopy result
  6. Covered by a Health Insurance System, which will cover colonoscopy as screening in patients with risk factors and alarm symptoms such as abdominal pain, change in stool texture, change in stool frequency, blood in stool/rectal bleeding, diarrhea, constipation, abdominal bloating, weight loss, tiredness.
* Control Group with risks and absence of polyps

  1. Signature of the informed consent indicating that the subject accepts to participate in the study and to comply with the requirements and restrictions inherent in this study.
  2. Subjects aged ≥18 years
  3. Otherwise healthy individuals with recognized risk factors for CRC development defined by either heredity and/or obesity and/or smoking and/or excess alcohol consumption and/or hyperlipidaemia.
  4. Subject be willing to undergo FOBT test, colonoscopy, and tissue biopsy
  5. Subject has negative CRC diagnosis according to colonoscopy result
  6. Covered by a Health Insurance System, which will cover colonoscopy as screening in patients with risk factors and alarm symptoms such as abdominal pain, change in stool texture, change in stool frequency, blood in stool/rectal bleeding, diarrhea, constipation, abdominal bloating, weight loss, tiredness.
* Control Group with no risks

  1. Signature of the informed consent indicating that the subject accepts to participate in the study and to comply with the requirements and restrictions inherent in this study.
  2. Subjects aged ≥40 years
  3. Otherwise healthy individuals without any recognized risk factors for CRC development defined by either heredity and/or obesity and/or smoking and/or excess alcohol consumption and/or hyperlipidemia.
  4. Subject be willing to undergo FOBT test
  5. Subject has negative FOBT result

Exclusion Criteria:

* For the CRC Group

  1. Legal incapacity or limited legal capacity
  2. Subject did not sign the Informed Consent form
  3. Subject who, according to the investigator's assessment, presents with an unstable medical condition contraindicating the performance of the planned blood test, stool test or breath test
  4. Subject has had surgery in the previous 6-8 weeks or is under medication for CRC treatment.
* For the control groups

  1. Legal incapacity or limited legal capacity
  2. Subject did not sign the Informed Consent form
  3. Previous history of any type of cancer
  4. Gastrointestinal disorders or other serious acute or chronic diseases

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects aged over 18 for all groups except the control group with no risk where in this group subjects are aged ≥ 40 years.
Sampling Method: Non-Probability Sample
Enrollment: 4100 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
ONCO CTC expression pattern of ONCOSCREEN tools in CRC patients and healthy controls using colonoscopy as the reference method. | At the day of visit/sampling and through study completion, an average of 3 years
  Blood samples will be collected to assess various novel biomarkers associated with CRC.
ONCO NMR expression pattern | At Day1 and through study completion, an average of 3 years
  Blood samples will be collected to assess various novel biomarkers associated with CRC.
ONCO CRISPR expression pattern | At Day1 and through study completion, an average of 3 years
  Blood and stool samples will be collected to assess various novel biomarkers associated with CRC.
ONCO VOC expression pattern | At Day1 and through study completion, an average of 3 years
  Breath samples will be collected to analyze volatile organic compounds (VOCs). By examining the electrochemical signal responses using pattern recognition algorithms, researchers can identify early indicators distinguishing between CRC-linked and healthy categories.
Evaluation of genetic risks associated to CRC | At Day1 and through study completion, an average of 3 years
  Buccal swabs will be collected to evaluate genetic risks associated to CRC. Analyzing buccal swab samples can identify genetic variations linked to an increased CRC risk, enhancing personalized screening accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: Markus MOELHER, MD, PhD, Principal Investigator — University Medical Center Mainz
Locations (8):
- Bulgaria (2):
  - Military Medical Academy Sofia, Gastroenterology Clinic, 3 Sveti Georgi Sofiiski str., Sofia 1606, Bulgaria, Sofia
  - University Specialised Hospital for Active Treatment of Oncology Departement of Gastroenterology., Sofia
- UFC: Université de Franche-Comté Oncology department CHU Besançon, Besançon, France
- Germany (2):
  - MKI UKSH Lübeck, Lübeck
  - UMC Mainz: University Medical Center Mainz, Mainz-GE
- LSMU: Lithuanian University of Health Sciences Gastroenterology Department,, Kaunas, Lithuania
- IPO: Instituto Português de Oncologia, Porto, Portugal
- IBO: Institutul Oncologic Prof. Dr. Alexandru Trestioreanu București, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website of the clinical study — https://oncoscreen.health/